CLINICAL TRIAL: NCT07044635
Title: Radiation Therapy in Reduced Dose and Hypofractionated Schedule After Trans-Oral Robotic Surgery in Intermediate Risk HPV-Mediated Oropharyngeal Squamous Cell Carcinoma
Brief Title: Shortened Course of Radiation Therapy After Trans-oral Robotic Surgery in Patients With HPV-Mediated Oropharyngeal Squamous Cell Carcinoma.
Acronym: RAD RAPTORS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI191152
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma; HPV-mediated Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 10 fractions of radiation therapy (Experimental)
  Interventions: Radiation: Radiation Therapy
- Radiation therapy with chemotherapy, if applicable, per standard of care (Active Comparator)
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Reduced dose and Hypofractionated radiation therapy

SUMMARY:
The goal of this study is to evaluate if a shorter course of therapy can improve the quality of life in patients receiving radiation therapy after trans-oral robotic surgery.

ELIGIBILITY:
Step 1 Registration: Pre-Operative Eligibility

Inclusion Criteria:

* Participant aged ≥ 18 years.
* Diagnosis of oropharyngeal squamous cell carcinoma.
* Eligible to receive transoral robotic surgery.
* P16 positivity or HPV positivity by in situ hybridization on pathological sampling of lymph node or primary oropharyngeal tumor.
* Pre-operative TTMV-HPV DNA test collected.

  * Standard of care tests completed within 60 days of registration may be used for screening.
  * Tests results are not required to confirm eligibility for step 1 registration.
* ECOG Performance Status ≤ 2
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* History of prior mucosal head and neck cancer treated with radiation therapy
* Prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of this study
* Participant has smoked cigarettes within 1 month of registration
* Prior systemic anti-cancer therapy or any investigational therapy ≤ 14 days or within five half-lives prior to starting study treatment, whichever is shorter.
* Known distant metastatic disease.
* Current evidence of any condition that would, in the Investigator's judgment, contraindicate the participant's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [participants may not receive the drug through a feeding tube], social/ psychological issues, etc.)
* Medical, psychiatric, cognitive, or other conditions that may compromise the participant's ability to understand the participant information, give informed consent, comply with the study protocol or complete the study.

Step 2 Registration - Experimental Arm

Inclusion Criteria:

* Completion of trans-oral robotic surgery.
* Pre- and post-operative TTMV-HPV DNA test results obtained.
* For participants of child bearing potential: Negative pregnancy test or evidence of permanent surgical sterilization. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution
  * ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year
* Participants of childbearing potential must agree to use a highly effective method of contraception as described in Section 5.5.2.

Exclusion Criteria:

* Meets ALL of the following criteria for low-risk disease (Note: participants may meet some without being excluded):

  * Pre-operative TTMV-HPV DNA positive
  * Post-operative TTMV-HPV DNA negative
  * Disease: pT1 with ≤ 1 lymph nodes OR pT2N0
  * <10 pack year smoking
  * No extranodal extension
  * Negative surgical margins
  * No perineural invasion
  * No lymphovascular invasion
* Meets ANY of the following criteria for high-risk:

  * Post-operative TTMV-HPV DNA positive
  * Surgical margin positive -->1 mm extranodal extension --≥ 5 lymph nodes
* Current evidence of any condition that would, in the Investigator's judgment, contraindicate the participant's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [participants may not receive the drug through a feeding tube], social/ psychological issues, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Stable or improved FACT-HN at 6 months post-treatment compared to baseline. | 2 years
  To evaluate if a shorter course of therapy can improve quality of life in patients receiving adjuvant radiation therapy after TORS.

SECONDARY OUTCOMES:
The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type. | 2 years
  To assess the safety and tolerability of reduced-dose adjuvant radiation therapy in the study population.
The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by severity (as defined by the NIH CTCAE, version 5.0). | 2 years
  To assess the safety and tolerability of reduced-dose adjuvant radiation therapy in the study population.
The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by seriousness. | 2 years
  To assess the safety and tolerability of reduced-dose adjuvant radiation therapy in the study population.
The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by duration. | 2 years
  To assess the safety and tolerability of reduced-dose adjuvant radiation therapy in the study population.
The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by relationship to study drug. | 2 years
  To assess the safety and tolerability of reduced-dose adjuvant radiation therapy in the study population.
Progression-free survival (PFS) as defined as the time from surgery to the time of recurrence or death from any cause. | 4 years
  To assess PFS at 1-year post-radiation.
Overall survival (OS) as defined as the time from registration until death from any cause. | 4 years
  To assess overall survival in this study population.
The proportion of participants who experience local-regional recurrence. | 4 years
  To assess the local-regional recurrence rate.
The proportion of participants who experience distant recurrence. | 4 years
  To assess the distant recurrence rate.
The proportion of participants who experience recurrence. | 4 years
  To assess the overall recurrence rate.
Stable or improved MDADI defined by patient quality of life. | 4 years
  To assess patient-reported quality of life.
Stable or improved FACT-HN at 12 months post-treatment compared to baseline. | 4 years
  To evaluate if a shorter course of therapy can improve quality of life in patients receiving adjuvant radiation therapy after TORS.
This endpoint is restricted to participants who are able to work prior to treatment. Of those participants, the proportion who remain able to work 6 months after treatment as assessed by the FACT-HN. | 4 years
  To evaluate the ability for participants to return to work after a shorter course of adjuvant radiation therapy following TORS.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States